CLINICAL TRIAL: NCT03973892
Title: Remote Brain Microhaemorrhages May Predict Haematoma in Glioma Patients Treated With Radiation Therapy
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: 29651771
Record Dates: First submitted 2019-05-31; First posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cere — Magnetic Rseonance imaging for brain tumour follow-up

SUMMARY:
the study aim to evaluate the prevalence of cerebral remote microhaemorrhages (RMH) and remote haematomas (RH) using magnetic resonance susceptibility-weighted imaging (SWI) among patients treated for gliomas during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* glioma

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with glioma and folllow up with magnetic resonance imaging
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
number of microhaemorrhages (RMH) on magnetic resonance imaging | one year
number of remote haematomas (RH) on magnetic resonance imaging | one year

IPD SHARING:
Plan to Share IPD: Undecided